CLINICAL TRIAL: NCT06718647
Title: Efficacy and Tolerability of Low-Dose Versus Standard-Dose Enzalutamide in Advance Prostate Cancer: a Real-World Evidence Study
Brief Title: Efficacy and Tolerability of Low-Dose Enzalutamide in Prostate Cancer
Acronym: LODE
Status: Not yet recruiting | Type: Observational
Sponsor: Monica Boitano (Other)
Responsible Party: Sponsor-Investigator, Monica Boitano, Scientific Coordinator, Ente Ospedaliero Ospedali Galliera
Organization: Ente Ospedaliero Ospedali Galliera (Other)
Other Study IDs: LODE
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer Metastatic Disease
Keywords: Enzalutamide; Low-Doses; Prostatic neoplasms; Elderly; Adverse event; Metastatic prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Low Dose of Enzalutamide: Low Dose of Enzalutamide: ≤ 50% of the standard dose
- Intermediate Dose of Enzalutamide: Intermediate Dose of Enzalutamide: > 50% and ≤ 80% of the standard dose
- High Dose of Enzalutamide: High Dose of Enzalutamide: > 80% of the standard dose

SUMMARY:
Prostate cancer is the most common cancer in men in the United States and the second leading cause of cancer-related mortality in males. Since 2014, its incidence has increased by 3% annually, primarily due to a rise in advanced-stage cases. In Italy, over 41.000 cases were diagnosed in 2023, with 8.200 deaths. Enzalutamide, an androgen receptor inhibitor, is effective in treating metastatic prostate cancer but often requires dose reductions to improve tolerability in frail patients. Recent studies have shown that lower doses (≤ 80 mg per day) can maintain efficacy while improving safety and tolerability, with outcomes comparable to the standard dose (160 mg per day) in terms of overall survival, progression-free survival, and prostate-specific antigen response.

Based on the results observed in these studies, the investigators expect that in our retrospective cohort of patients with metastatic prostate cancer, those who received low doses of enzalutamide will have a 1 year progression-free survival comparable to the full dose. The investigators will also expect a lower rate of adverse events.

DETAILED DESCRIPTION:
Prostate cancer is the most frequent cancer in males in the United States, with 299.000 new cases estimated in 2024, and it is the second leading cause of cancer-related death in men. Since 2014, the prostate cancer incidence rate has risen by 3% per year, mostly driven by 4-5% per year increases for regional-stage and distant-stage diagnoses that began as early as 2011. Localized-stage disease also increased from 73.5 per 100.000 in 2014 to 84.8 per 100.000 in 2019, although the trend is not yet statistically significant. A recent study estimated that more than one half of men in the United States living with metastatic prostate cancer were initially diagnosed with localized or regional stage disease. In Italy, there were more than 41.000 diagnosed cases in 2023 and 8.200 deaths, accounting for nearly one-fifth of all cancers detected in men, and over 560.000 prevalent cases of men living with prostate.

Enzalutamide is a new generation oral androgen-receptor selective inhibitor that induces tumor regression and growth suppression in patients with metastatic prostate cancer. It is effective and well tolerated, compared with other anticancer drugs (ex-chemotherapy), but in real practice, very often in patients with comorbidity or poor performance status is necessary reduce the dose to reduce fatigue or other adverse events.

The standard recommended dosage of 160 mg per day has multiple side effects and dose reductions are often required.

Several randomized studies have underscored the importance of enzalutamide in treating prostate cancer. Initially approved by the Food and Drug Administration in 2012 for patients with metastatic castration-resistant prostate cancer who had previously received docetaxel, its indications were updated in October 2020 to include patients with castration-resistant prostate cancer experiencing biochemical relapse, or with metastatic castration-sensitive prostate cancer.

In phase I study enzalutamide (MDV3100) was administered with dose between 30 and 600 mg per day. There was a linear increase in steady state serum concentration with dose, but antitumor effects were observed at all doses, including 40-60 mg per day. The severity of treatment related adverse effects including fatigue and neurological disorders was associated with drug dose.

Recent data suggest its efficacy may be retained at lower doses with significant improvement in safety and tolerability. In two previously observational studies, in metastatic prostate cancer low-dose enzalutamide (≤ 80 mg per day) compared to standard dose (160 mg per day) did not show difference in overall survival and prostate-specific antigen progression-free survival. Interestingly, there was a trend towards a better prostate-specific antigen response and a significantly longer life among the low-dose group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological diagnosis metastatic prostate cancer;
* Enzalutamide therapy taken between 01/08/2014 and 31/12/2023;
* Age ≥ 18 years;
* Signed Informed consent.

Exclusion Criteria:

* Clinically significant cardiovascular disease for example cerebrovascular accidents (<=6 months), myocardial infarction (<=3 months), unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure (CHF); uncontrolled hypertension or bradycardia
* Patients who died within one month of starting treatment with Enzalutamide for all causes;
* Uncontrolled concomitant diseases.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of male patients aged 18 years or older with a histopathological diagnosis of metastatic prostate cancer who received Enzalutamide between 01/08/2014 and 31/12/2023.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 1 year
  The primary objective of this retrospective observational study is to evaluate whether low or intermediate doses of enzalutamide are comparable to the full dose in terms of 1-year average progression free survival time from the start of treatment, considering the event as the pathological progression of the disease.
Adverse events | At end of treatment with Enzalutamide
  To evaluate the rate of adverse events worsening between low, intermediate and full dose groups. As adverse events, fatigue, hypertension and neurological disorders will be assessed as adverse events of special interest.

SECONDARY OUTCOMES:
Overall Survival | 1 year
  To evaluate the Overall Survival, in terms of 1 year average survival time from the start of treatment, between low or intermediate doses compared to full dose;
Overall Survival | 3 years
  To evaluate the Overall Survival (OS), in terms of 3-years average survival time from the start of treatment, between low or intermediate doses compared to full dose;
Prostate Specific Antigen response | 3 months
  To evaluate the Prostate Specific Antigen response at 12 weeks between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea De Censi, Study Chair — Ente Ospedaliero Ospedali Galliera
Locations (1):
- Ente Ospedaliero Ospedali Galliera, Genoa, GENOA, Italy

IPD SHARING:
Plan to Share IPD: No